CLINICAL TRIAL: NCT06435585
Title: Responders and Non-responders in the Management of Heart Failure - Significance of Genetic Influence and Identification of Novel Informative Biomarkers
Acronym: Responders
Status: Recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Camilla Hage, Associate Professor, Karolinska University Hospital
Other Study IDs: 218/443-31
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Pathophysiology
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, whole blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A biobank within the Swedish national heart failure quality registry SwedeHF.

DETAILED DESCRIPTION:
The national heart failure quality registry SwedeHF started in 2003. It is the world's largest continuous HF registry enrolling clinician-judged HF (regardless of LVEF) at time of hospital or clinical visit. Eighty variables are entered into an electronic database managed by the Uppsala Clinical Research Center (UCR). There are >140,000 registrations from >110,000 unique patients from 70 hospitals in Sweden.

University hospitals in Sweden with access to central biobanking will collect a high-quality biobank linked to SwedeHF consisting of blood plasma, whole blood and urine enabling genetic, proteomic and metabolomic analyses as well as analyses of different biomarkers of interest for HF patients. This will provide unique opportunities for future research within the national SwedeHF registry.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Heart failure defined by symptoms and signs of heart failure as judged by the local investigator
3. Registered in SwedeHF

Exclusion Criteria:

1. Plasma donation within 1 month of enrolment or any blood donation/blood loss >500 mL during the 3 months prior to enrolment
2. Previous allogeneic bone marrow transplant (genetics)
3. In the opinion of the investigator, condition/s that may either put the patient at risk on participation or influence the results or the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAtients with heart failure in Sweden with a registration in SwedeHF.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify responders to guideline-directed medical therapy | 2 and 5 years
  To identify which patient will be a non-responder resulting in a poor outcome, despite being on recommended treatment according to guidelines.
Differences in morbidity between responders and non-responders to guideline-directed medical therapy | 2 years
  To characterize differences between responders and non-responders in terms of morbidity after 2-years follow-up.
Differences in mortality between responders and non-responders to guideline-directed medical therapy | 2 years
  To characterize differences between responders and non-responders in terms of mortality after 2-years follow-up.
Predictors of responders and non-responders to guideline-directed medical therapy | 2 and 5 years
  To integrate information regarding clinical characteristics, diagnostic markers and genetics to determine underlying mechanisms behind different responses to treatment.

SECONDARY OUTCOMES:
Differences between responders and non-responders regarding mortality | 2 and 5 years
  To evaluate the differences between HFrEF and HFpEF patients in terms of mortality and after 2 and 5 years follow-up, respectively.
Differences between responders and non-responders regarding morbidity | 2 and 5 years
  o evaluate the differences between HFrEF and HFpEF patients in terms of morbidity after 2 and 5 years follow-up, respectively.
Predictors of mortality in responders and non-responders | 2 and 5 years
  To evaluate the differences in mortality between patients with HFrEF and HFpEF by integrating information from clinical characteristics, diagnostic markers and genetics in order to have a further understanding of the underlying pathophysiology involved in HF development and prognosis with the aim to facilitate improved individualized therapy with less adverse effects and to identify novel treatment targets.
Predictors of morbidity in responders and non-responders | 2 and 5 years
  To evaluate the differences in morbidity between patients with HFrEF and HFpEF by integrating information from clinical characteristics, diagnostic markers and genetics in order to have a further understanding of the underlying pathophysiology involved in HF development and prognosis with the aim to facilitate improved individualized therapy with less adverse effects and to identify novel treatment targets.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will only be within investigators. Beyond study investigators data sharing requires new ethical approval.